CLINICAL TRIAL: NCT03461354
Title: Phase II Randomized Trial of an Oral Formulation Containing a Mucoadhesive Polymer Hydrogel Vehicle (MucoLox®) to Mitigate Mucositis Symptoms in Head/Neck Cancer Patients Receiving Radiation ± Chemotherapy
Brief Title: MucoLox Formulation to Mitigate Mucositis Symptoms in Head/Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis indicated study closure
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Professional Compounding Centers of America (Industry); Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00081365; 00024266 (Other: Advarra IRB); LCI-HN-MUC-LOX-001 (Other: Atrium Health)
Record Dates: First submitted 2018-02-27; First posted 2018-03-12 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Mucositis Oral; Head and Neck Cancer
Keywords: Oral rinse; Chemotherapy and Radiation Side Effects
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Mucolox Arm
  Interventions: Other: MucoLox
- B (Active Comparator): Sodium Bicarb Control Arm
  Interventions: Other: Sodium Bicarbonate

INTERVENTIONS:
Other: MucoLox — MucoLox formulation, with MucoLox as the delivery vehicle, combined with preserved water, beta-glucan, dexpanthenol, and glutamine
  Arms: A
Other: Sodium Bicarbonate — Sodium bicarbonate oral rinse
  Arms: B

SUMMARY:
This study will examine if the administration of prophylactic MucoLox formulation versus sodium bicarbonate mouthwash in subjects with head/neck cancer receiving radiation ± chemotherapy will result in significantly fewer subjects experiencing severe mucositis.

DETAILED DESCRIPTION:
The primary objective of this double-arm, single-blinded, Phase II randomized study is to compare the area under the curve (AUC) for the Oral Mucositis Daily Questionnaire (OMDQ) mouth and throat soreness (MTS) question 2 (Q2) score over a one-month period in subjects receiving the MucoLox formulation versus sodium bicarbonate rinse (as the control) for the prevention of severe mucositis in subjects with head/neck cancer receiving radiation ± chemotherapy. Secondary objectives include comparing the time to OMDQ MTS Q2 > 2 between the two arms; estimating and comparing opioid use defined as the average morphine equivalent daily dose (MEDD) at each clinic visit; assessing and comparing changes in the remaining OMDQ questions longitudinally throughout study; evaluating and comparing the duration of symptom relief in those who experience any degree of oral mucositis; evaluating and comparing the frequency of delays in [chemotherapy and/or radiation] therapy throughout the study period; and summarizing and comparing the prevalence and grade of oral mucositis at each clinic visit. The safety objective is to summarize the rates of potential side effects related to each oral formulation. A total of 60 eligible subjects will be enrolled and randomized in a 1:1 fashion to one of the treatment arms. Subjects on the control arm (sodium bicarbonate) who experience severe mucositis will have the option to crossover to the Mucolox arm for an additional 7 ± 2 days or until day 29 ± 5 days, whichever is longer.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria:

1. Confirmed head/neck cancer scheduled to receive at least a 28-day course of radiation to the head/neck area (radiation field must include at least one mucosal site within the oral cavity space, oropharynx, hypopharynx or larynx). Subjects must be planned to receive a minimum cumulative dose of 40 Gy and maximum dose of 72 Gy of radiation. Subjects may or may not be scheduled to receive concomitant platinum-based chemotherapy administered with radiation
2. At least 18 years of age
3. ECOG performance status less than or equal to 2 or Karnofsky performance score greater than or equal to 70%.
4. Able and willing to complete OMDQ as determined by the treating Investigator
5. Able and willing to swish/spit the oral formulation as determined by the treating Investigator
6. Able and willing to provide informed consent

Exclusion Criteria

Subjects must not meet any of the following criteria:

1. Receiving any other pharmacological treatment within 1 week of initiation of study treatment for oral mucositis, excluding analgesics, antibiotics, antifungals, and hydration for symptom management. Subjects must also agree to not use any other mouthwash formulations to prevent or treat mucositis during the course of the study.

   1. The subject's enrolling investigator must agree to not prescribe any other mouthwash formulations to prevent or treat oral mucositis during protocol-directed treatment (Note: subjects may receive standard of care treatment if the subject develops oral mucositis and discontinues study treatment [or may crossover to Arm A if randomized to Arm B]).
   2. Subjects must also agree to not use any other mouthwash formulations to prevent or treat oral mucositis during protocol-defined treatment.

   i. Agents suggested to modify oral mucositis risk or course that are not allowed include sodium bicarbonate, magic mouthwash formulations, amifostine, benzydamine, cevimeline, glutamine rinse, topical GM-CSF, interleukin-11, chlorhexidine, hydrogen peroxide, diphenhydramine, palifermin, pilocarpine, steroid rinses, sucralfate, and various oral rinse medical devices
2. Untreated or unresolved oral infections, including oral candidiasis or active lesions due to oral herpes simplex virus infection that in the opinion of the investigator would compromise study outcomes.
3. Signs and symptoms of any mouth and/or throat condition or active dental disease that would impair the ability to administer the mouthwash and/or assess the development of oral mucositis, as determined by the Investigator.
4. Presence of baseline grade > 1 oral mucositis per WHO criteria as determined by the treating investigator
5. Receiving chronic immunosuppression as determined by the Investigator
6. Known hypersensitivity to any ingredients in the mouthwash formulations that may result in anaphylaxis.
7. Use, or suspicion of use, of illicit drugs or substances (self-reported) that may, in the opinion of the Investigator, have a reasonable chance of contributing to non-compliance, opioid abuse, drug toxicity, and/or otherwise skewing the trial result

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
AUC for the Oral Mucositis Daily Questionnaire mouth and throat soreness question #2 | One month
  To compare the area under the curve (AUC) for the Oral Mucositis Daily Questionnaire (OMDQ) mouth and throat soreness (MTS) question 2 (Q2) score over a one-month period in subjects receiving the MucoLox formulation versus sodium bicarbonate rinse (as the control) for the prevention of severe mucositis in subjects with head/neck cancer receiving radiation ± chemotherapy

SECONDARY OUTCOMES:
Time to OMDQ MTS > 2 | One month
  To compare the time to OMDQ MTS Q2 > 2 between the two arms
Opioid use (morphine equivalent daily dose) | Weekly during the one-month study period
  To estimate opioid use defined as the average morphine equivalent daily dose (MEDD) at each clinic visit: baseline, day 8 ± 2, day 15 ± 2, day 22 ± 2, and the final study visit (day 29 ± 5) and compare between the two arms
Assess remaining OMDQ questions | One month
  To assess changes in the remaining OMDQ questions longitudinally throughout study treatment and compare between the two arms.
Duration of symptom relief | One month
  To evaluate and compare the duration of symptom relief in those who experience any degree of oral mucositis between the two arms
Frequency of chemoradiation delays | One month
  To evaluate the frequency of delays in [chemotherapy and/or radiation] therapy throughout the study period and compare between the two arms.
Oral mucositis grade | Weekly during the one month study period
  To summarize the prevalence and grade of oral mucositis at each clinic visit: baseline, day 8 ± 2, day 15 ± 2, day 22 ± 2, and the final study visit (day 29 ± 5), as assessed by the treating investigator using the WHO criteria for grading, and compare between the two arms.
Comparison of self-reported OMDQ scores versus investigator-assessed mucositis | Weekly during the one month study period
  The Generalized McNemar's test will be used to analyze correlation between patient report OMDQ Q2 scores and oral mucositis grading assessed by treating investigator using WHO criteria.

OTHER OUTCOMES:
Drug-related adverse events | One month
  To summarize the rates of potential side effects related to each oral formulation, including but not limited to mouth discomfort, allergic reactions, exacerbation of mucositis symptoms, mouth ulcers, dry mouth, unpleasant taste or dysgeusia. Safety variables include AEs and SAEs related to the study treatment. Adverse events will be evaluated continuously throughout the study. Safety, tolerability, relationship to study treatment, and intensity will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Jai Patel, PharmD, BCOP, Principal Investigator — Levine Cancer Institute, Atrium Health (formerly Carolinas HealthCare System)
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT03461354/ICF_000.pdf